CLINICAL TRIAL: NCT04572685
Title: A Randomized, Open-Label, Parallel, Single-Dose Study to Evaluate the Pharmacokinetic Characteristics of LY03010 Process 1 and Process 2 Drug Product Versus INVEGA SUSTENNA After Intramuscular Injection in Schizophrenia Patients
Brief Title: Evaluate the PK of LY03010 Process 1 and Process 2 Drug Product vs INVEGA SUSTENNA After Intramuscular Injection in Schizophrenia Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Luye Pharma Group Ltd. (Industry)
Collaborators: Alliance for Clinical Trials in Oncology (Other); Evolution Research Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LY03010/CT-USA-102
Record Dates: First submitted 2020-05-08; First posted 2020-10-01 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Schizophrenia Patients
MeSH Terms: interventions — Paliperidone Palmitate

STUDY DESIGN:
Intervention Model Description: A single dose study in three parallel dosing groups of schizophrenia patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- LY03010 Process 1 (Experimental): Drug Product of Process 1 ( P1): 156 mg/vial; Single Injection on Day 1 during the entire 120 Day's study.
  LY03010 P1 using a non-sterile Active Pharmaceutical Ingredients (API) with an absolute ethanol recrystallization was manufactured by an optimized production process
  Interventions: Drug: Paliperidone Palmitate
- LY03010 Process 2 (Experimental): Drug Product of Process 2 (P2): 156 mg/vial; Single Injection on Day 1 during the entire 120 Day's study.
  LY03010 P2 using a sterile Active Pharmaceutical Ingredients (API) with an isopropanol recrystallization was manufactured by the same optimized production process as that used in P1.
  Interventions: Drug: Paliperidone Palmitate
- INVEGA SUSTENNA (Experimental): INVEGA SUSTENNA 156 mg/vial; Single Injection on Day 1 during the entire 120 Day's study
  Interventions: Drug: Paliperidone Palmitate

INTERVENTIONS:
Drug: Paliperidone Palmitate — A long acting extended release injectable suspension intended for monthly intramuscular administration
  Other Names: Paliperidone Injectable Product

SUMMARY:
The primary objectives of the study are to characterize the pharmacokinetic (PK) profiles of paliperidone in LY03010 P1 and P2 following a single IM injection in schizophrenia patients and to compare the PK of LY03010 P1 and P2 with that of INVEGA SUSTENNA® following a single IM injection of 156 mg dosage level.

DETAILED DESCRIPTION:
This is a randomized, open-label, parallel-group, single-dose study. Patients will undergo screening evaluations to determine eligibility within 28 days prior to study drug administration. About 36 patients will be randomized in a 1:1:1 ratio to 1 of 3 treatment groups. Patients will be admitted to the clinical facility the day before dosing (Day 0) and will be receiving an IM injection of study drug and completing the assigned study activity including PK sample collection on Day 1. Patients will be discharged on Day 2 after PK collection. All patients will return to the clinical site at designated study days for PK sample collections and assigned clinical procedures. End of study evaluation will be completed on Day 120.

Pharmacokinetics of the study medication will be assessed as primary outcome. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥18 to ≤65 years of age who meets diagnostic criteria for schizophrenia according to the Diagnostic and Statistical Manual of Mental Disorders Fifth Edition (DSM-V) for at least 1 year before screening
* Have been on a stable dose of oral antipsychotic medication(s) other than risperidone, paliperidone, clozapine, ziprasidone, or thioridazine for at least 4 weeks prior to screening
* Clinically stable based on clinical assessments and a Positive and Negative Syndrome Scale (PANSS) total score ≤70 as well as a PANSS HATE (hostility, anxiety, tension and excitement) subtotal score <16 at screening
* Clinical Global Impression-Severity (CGI-S) score of 1 to 4, inclusive
* Body mass index (BMI) ≥17.0 and ≤37kg/m2; body weight ≥50 kg
* Creatinine level within the normal range
* All female patients (childbearing potential and non-childbearing potential) must have a negative pregnancy test result at both screening and baseline.
* Sexually active fertile male patients must be willing to use acceptable contraception methods (such as double barrier methods of a combination of male condom with either cap, diaphragm or sponge with spermicide) from study drug dosing, throughout the study, and for another 80 days after the EOT visit (or at least 200 days after the dose, whichever is longer) if their partners are women of childbearing potential.

Exclusion Criteria:

* Primary and active DSM-V Axis I diagnosis other than schizophrenia
* Patients who meet DSM-V criteria for substance abuse (moderate or severe) with the exception of caffeine or nicotine in the past 6 months prior to screening, or test positive for barbiturate or alcohol at screening or baseline
* Patients who received any of following treatment:

  * Use of oral risperidone or paliperidone within 2 weeks before screening.
  * Use of clozapine, thioridazine or ziprasidone within 4 weeks before screening.
  * Use of 2-week depot formulation of risperidone within 3 months, 1-month depot formulation of risperidone or 9-hydroxy risperidone (INVEGA SUSTENNA) within 1 year,
* Known or suspected hypersensitivity or intolerance of risperidone, paliperidone, or any of their excipients (oral risperidone tolerability test should be completed during the screening period
* QTcF interval greater than 450 msec for males and 470 msec for females or a prior history or presence of circumstances
* Medical history (within 2 years) of clinically significant, gastrointestinal, cardiovascular, cerebrovascular, musculoskeletal, endocrine, hematologic, renal, hepatic, bronchopulmonary, neurologic, immunologic disorders, or drug hypersensitivity which, in the judgement of the Investigator, would interfere with the patient's ability to participate in the study
* History of dementia-related psychosis or Parkinson's Disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-01-22 (Actual); Primary Completion 2020-06-26 (Actual); Study Completion 2020-08-20 (Actual)

PRIMARY OUTCOMES:
To characterize the Maximum Plasma Concentration [Cmax]of LY03010 P1, P2 and INVEGA SUSTENNA following a single IM injection of 156 mg dosage level in schizophrenia patients | 120-Day
  The Cmax of LY03010 P1, P2 and INVEGA SUSTENNA will be measured
To characterize Area under the plasma concentration versus time curve (AUC) of LY03010 P1 and P2 and INVEGA SUSTENNA following a single IM injection of 156 mg dosage level in schizophrenia patients. | 120-Day
  The AUCs of LY03010 P1, P2 and INVEGA SUSTENNA will be evaluated
To compare the Cmax of LY03010 P1 and P2 with the Cmax of INVEGA SUSTENNA | 120-Day
  The relative bioavailability of LY03010 P1 and P2 to Invega Sustenna will be assessed
To compare the AUCs of LY03010 P1 and P2 with the AUCs of INVEGA SUSTENNA | 120-Day
  The relative bioavailability of LY03010 P1 and P2 to Invega Sustenna will be assessed

SECONDARY OUTCOMES:
To evaluate the safety and tolerability of tested drugs. Safety assessments include Incidence of adverse events. | 120 day
  AE will be monitored throughout of the study course
To evaluate the safety of the tested drugs-- Incident of abnormal vital sign | 120 Day
  Vital Sign will be measured on Day1 ,2, 4, 6, 8,10,12,15, 17,19, 22 ,29, 64, 92 and Day 120
To evaluate the safety of the tested drugs-- Incident of abnormal ECG Findings | 120 Day
  12-Lead ECG will be measured on Day 0, 29, 64, 92 and Day 120
To evaluate any abnormal movement symptoms measured by Abnormal Involuntary Movement Scale (AIMS). AIMS measures movement of each part of body muscle with score range of 0-4, 0 means None and 4 means Severe. | 120-Day
  AIMS will be measured on Day 0, 15, 29, 64, 92 and Day 120
To evaluate any abnormal movement symptoms measured by Barnes Akathisia Rating Scale (BARS). BARS is a rating scale for drug-induced akathisia with a range of 0-14; 0 means Normal and 14 means Severe. | 120-Day
  BARS will be measured on Day 0, 15, 29, 64, 92 and Day 120
To evaluate any suicidal attempts measured by Columbia Suicide Severity Rating Scale ( C-SRRS). C-SRRS measures the suicidal intensity of ideation and attempt with score of 1-5; 1 means the least severe and 5 means the most severe. | 120-Day
  C-SSRS will be measured on Day 0, 29, 64, 92 and Day 120

CONTACTS AND LOCATIONS:
Overall Officials: Luye Pharma, Study Chair — Luye Pharma Group
Locations (1):
- Hassman Research Institute, Berlin, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No